CLINICAL TRIAL: NCT02056990
Title: Screening of Athletes for Prevention of Injury and Optimisation of Performance
Brief Title: Screening of Athletes
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. F. Staes, Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56252
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Individual Differences; Motor Activities
Keywords: Athletes
MeSH Terms: conditions — Motor Activity | interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- training advise
  Interventions: Other: Advice

INTERVENTIONS:
Other: Advice

SUMMARY:
Athletes have to participate in screenings in order to reduce injuries. Up-to-now most screenings are purely clinically based. Literature, however, indicates the importance of knowledge on deviant movement patterns as possible risk factors for injuries. From this perspective, the current project aims to measure movement patterns, gait and running in young athletes to optimise training and prevent injuries.

2D- and 3d registration methods, force plate data and pressure plate data will be used to document the performance of the athletes.

ELIGIBILITY:
Inclusion Criteria:

1. Selected by the Flemish Athletics League
2. Level: B1, B2 en C
3. Age categories: 16-22 years
4. No injuries at lower back and lower extremities in the past 6 months
5. Signing informed consent

Exclusion Criteria:

1. Not selected by the Flemish Athletics League
2. Injuries at lower quadrant

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes will be selected from a list offered by the Flemish Atlethics League. This incorporates a group of athletes with potential to become Elite Athletes of the highest international level
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Kinematic and kinetic data | March - June 2014 (3 months)
  Angles at different joints will be investigated with 3D movement analysis methods. Kinetic data (joint moments) will be calculated with 3D movement analysis methods.
  Center of pressure measures will be calculated on the basis of force plate data.
  Gait, running, jumps, postural balance will be investigated. Plantar pressure parameters will be calculated on the basis of plantar pressure measurements.

SECONDARY OUTCOMES:
2 D parameters | March - June 2014 (3 months)
  Video analysis methods (Dartfish) will be used to calculate joint angles during jumps

OTHER OUTCOMES:
Sports activities,personal demographics, injury history | March - June 2014 (3 months)
  Sports activities, personal demographics and injury history will be documented through existing information from the medical department (Physical Rehabilitation of University Hospitals Leuven)

CONTACTS AND LOCATIONS:
Overall Officials: Filip F Staes, Professor, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/UZLeuven, Leuven, Vlaams-Brabant, Belgium